CLINICAL TRIAL: NCT00117403
Title: Evaluation of the Safety, Tolerability and Impact on Biomarkers of Anti-Oxidant Treatment of Mild to Moderate Alzheimer's Disease
Brief Title: Anti-Oxidant Treatment of Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Collaborators: Alzheimer's Disease Cooperative Study (ADCS) (Other)
Responsible Party: Paul Aisen, MD, Alzheimer's Disease Cooperative Study
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IA0067
Record Dates: First submitted 2005-06-30; First posted 2005-07-06 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Alzheimer's Disease
Keywords: dementia; anti-oxidant; biomarkers; alpha-tocopherol; CoQ
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Vitamin E; Ascorbic Acid; Thioctic Acid; Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): vitamin E 800 IU, vitamin C 200 mg, and alpha-lipoic acid 600 mg formulated into three capsules, one capsule given three times per day with meals, plus two placebo wafers three times per day with meals
  Interventions: Drug: Vitamin E, Vitamin C, and Alpha-lipoic Acid; Drug: Placebo wafers
- 2 (Experimental): CoQ 400 mg, compounded as a wafer, two wafers three times per day with meals, plus one placebo capsule three times per day with meals
  Interventions: Drug: Coenzyme Q; Drug: Placebo capsules
- 3 (Placebo Comparator): two placebo wafers three times per day with meals, plus one placebo capsule three times per day with meals
  Interventions: Drug: Placebo capsules; Drug: Placebo wafers

INTERVENTIONS:
Drug: Vitamin E, Vitamin C, and Alpha-lipoic Acid — vitamin E 800 IU, vitamin C 200 mg, and alpha-lipoic acid 600 mg formulated into three capsules, one capsule given three times per day with meals
  Arms: 1
Drug: Coenzyme Q — 400 mg, compounded as a wafer, two wafers three times per day with meals
  Arms: 2
Drug: Placebo capsules — one placebo capsule three times per day with meals
  Arms: 2; 3
Drug: Placebo wafers — two placebo wafers three times per day with meals
  Arms: 1; 3

SUMMARY:
The purpose of this study is to examine the safety and effectiveness of two anti-oxidant treatment regimens in patients with mild to moderate Alzheimer's disease. The anti-oxidant treatments include vitamin E + C + alpha-lipoic acid, and Coenzyme Q (CoQ).

DETAILED DESCRIPTION:
Oxidative damage has been shown to be a factor in Alzheimer's disease (AD), and some studies have suggested that supplemental anti-oxidants can decrease the risk of AD or slow its progression. There are many candidate antioxidants, including combinations, which could be neuroprotective in established AD or could have efficacy in the prevention of AD. However, testing each of the possibilities in standard clinical trials is prohibitively expensive. This study will examine antioxidant supplements or vitamins which target specific cellular compartments, and look for evidence of biologically relevant effects in AD by measurement of biomarkers in CSF.

Two general cellular compartments where antioxidant supplements may act are the cytosol and mitochondria. The study will examine a combination of antioxidants that act primarily at cytosolic sites (vitamin E + C + α-lipoic acid) and a single mitochondrial antioxidant, coenzyme Q10.

This multicenter trial will recruit 75 participants who will be randomized into three groups:

1. 25 participants will be given a combination of vitamin E 800 IU, vitamin C 200 mg, and alpha-lipoic acid 600 mg formulated into three capsules, one capsule given three times per day with meals, plus two placebo wafers three times per day with meals;
2. 25 participants will be given CoQ 400 mg, compounded as a wafer, two wafers three times per day with meals, plus one placebo capsule three times per day with meals;
3. 25 participants will be given both the placebo wafers, two wafers three times per day with meals, plus one placebo capsule three times per day with meals.

The treatment period will last four months. The effects of the two anti-oxidant treatments will be evaluated by measuring biomarkers in blood and cerebrospinal fluid (CSF) at the beginning and end of the 4-month period.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged 60-85, inclusive
* Diagnosis of probable Alzheimer's disease
* English-speaking; Spanish-speaking if individual site allows
* Study partner or caregiver to assure compliance
* Mini-Mental State Examination score at screening visit greater than 14
* Female participants either surgically sterile or postmenopausal for over 1 year
* Stable medical condition for 3 months prior to screening, with no significant abnormal liver, kidney, or blood studies
* Stable medications for 4 weeks prior to screening
* Able to take oral medications
* Modified Hachinski Ischemic Index less than or equal to 4
* CT or MRI since onset of memory impairment demonstrating the absence of a clinically significant focal lesion
* Physically acceptable for this study as confirmed by medical history, physical exam, neurological exam, and clinical tests

Exclusion Criteria:

* Significant neurologic disease such as Parkinson's disease, stroke, brain tumor, multiple sclerosis, or seizure disorder
* Major depression in the past 12 months, major mental illness such as schizophrenia, or recent (in past 12 months) alcohol or substance abuse
* History of invasive cancer within the past two years (excluding non-melanoma skin cancer)
* Contra-indications to lumbar puncture
* Use of any investigational agents within 30 days prior to screening
* Major surgery within 8 weeks prior to the Baseline Visit
* Uncontrolled cardiac conditions or severe unstable medical illnesses
* Antiretroviral therapy for human immunodeficiency virus (HIV)
* Conditions that will contribute to oxidative stress: current cigarette or cigar smokers (within past month), diabetics on insulin or poorly controlled on oral hypoglycemics
* Residence in skilled nursing facility
* Blindness, deafness, language difficulties or any other disability which may prevent the participant from participating or cooperating in the protocol

Note: Exceptions to these criteria may be considered on a case-by-case basis, at the discretion of the Project Director.

Excluded Medications:

* Experimental drugs
* Coumadin
* Insulin
* Immunosuppressive agents: prednisone and other corticosteroids (taken orally or by injection), methotrexate, cyclophosphamide, cyclosporin, tacrolimus, etc.
* HIV protease inhibitors
* Neuroleptics and lithium
* Anti-cancer agents (exception: stable doses of hormonal therapy, e.g. Lupron, estrogen, are permitted)

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2006-01; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
effect on cerebrospinal fluid (CSF) biomarkers related to oxidative damage | baseline and 4 months

SECONDARY OUTCOMES:
change in plasma and CSF concentrations of a-beta42 and a-beta40 | baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Galasko, MD, Principal Investigator — University of California, San Diego
Locations (13):
- United States (13):
  - University of Arizona, Tucson, Arizona
  - University of California- Irvine, Irvine, California
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - Wien Center, Mount Sinai Medical Center, Miami Beach, Florida
  - University of Kentucky, Lexington, Kentucky
  - University of Medicine and Dentistry of New Jersey, Piscataway, New Jersey
  - Neurological Care of CNY, Syracuse, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, North Charleston, South Carolina
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Sano M, Ernesto C, Thomas RG, Klauber MR, Schafer K, Grundman M, Woodbury P, Growdon J, Cotman CW, Pfeiffer E, Schneider LS, Thal LJ. A controlled trial of selegiline, alpha-tocopherol, or both as treatment for Alzheimer's disease. The Alzheimer's Disease Cooperative Study. N Engl J Med. 1997 Apr 24;336(17):1216-22. doi: 10.1056/NEJM199704243361704. PMID 9110909
- [Background] Behl C. Alzheimer's disease and oxidative stress: implications for novel therapeutic approaches. Prog Neurobiol. 1999 Feb;57(3):301-23. doi: 10.1016/s0301-0082(98)00055-0. PMID 10096843
- [Background] Zandi PP, Anthony JC, Khachaturian AS, Stone SV, Gustafson D, Tschanz JT, Norton MC, Welsh-Bohmer KA, Breitner JC; Cache County Study Group. Reduced risk of Alzheimer disease in users of antioxidant vitamin supplements: the Cache County Study. Arch Neurol. 2004 Jan;61(1):82-8. doi: 10.1001/archneur.61.1.82. PMID 14732624
- [Derived] Galasko DR, Peskind E, Clark CM, Quinn JF, Ringman JM, Jicha GA, Cotman C, Cottrell B, Montine TJ, Thomas RG, Aisen P; Alzheimer's Disease Cooperative Study. Antioxidants for Alzheimer disease: a randomized clinical trial with cerebrospinal fluid biomarker measures. Arch Neurol. 2012 Jul;69(7):836-41. doi: 10.1001/archneurol.2012.85. PMID 22431837